CLINICAL TRIAL: NCT03042611
Title: A Prospective, Randomized, Double-Blinded, Placebo-Controlled, Multinational, Multicenter, Parallel-group, Phase III Study to Evaluate the Efficacy and Safety of Apatinib Plus Best Supportive Care (BSC) Compared to Placebo Plus BSC in Patients With Advanced or Metastatic Gastric Cancer
Brief Title: A Study to Evaluate Rivoceranib Plus Best Supportive Care Compared to Placebo Plus Best Supportive Care in Participants With Gastric Cancer
Acronym: ANGEL
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Elevar Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: LSK-AM301
Record Dates: First submitted 2017-01-24; First posted 2017-02-03 (Estimated); Results first posted 2022-07-08 (Actual); Last update posted 2022-07-08 (Actual); Status verified 2022-06

CONDITIONS: Gastric Cancer; Gastric Adenocarcinoma
Keywords: Gastric Cancer; Gastric Adenocarcinoma; Gastro-esophageal Cancer; Gastro-esophageal Junction Cancer; Stomach Cancer; Tumor; Oncology; Antiangiogenesis; Metastatic
MeSH Terms: conditions — Stomach Neoplasms; Neoplasms; Neoplasm Metastasis | interventions — apatinib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Rivoceranib Plus BSC (Experimental): Participants will receive rivoceranib 700 milligrams (mg) orally once per day during each cycle plus BSC. BSC is defined as palliative, non-cancer therapy. Each cycle duration is 28 days.
  Interventions: Drug: Rivoceranib
- Placebo (Experimental): Participants will receive matching placebo to rivoceranib orally once per day during each cycle plus BSC. BSC is defined as palliative, non-cancer therapy. Each cycle duration is 28 days.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Rivoceranib — Oral tablet
  Other Names: Apatinib
  Arms: Rivoceranib Plus BSC
Drug: Placebo — Oral tablet
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of rivoceranib plus best supportive care (BSC) compared to placebo plus BSC in participants with advanced or metastatic gastric cancer (GC).

ELIGIBILITY:
Inclusion Criteria:

1. Documented primary diagnosis of histologic- or cytologic-confirmed adenocarcinoma of the stomach or gastroesophageal junction.
2. Locally advanced unresectable or metastatic disease that has progressed since last treatment.
3. One or more measurable or nonmeasurable evaluable lesions per Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST 1.1).
4. Failure or intolerance to at least 2 prior lines of standard chemotherapies with each containing one or more of the following agents:

   * fluoropyrimidine (intravenous [IV] 5-fluorouracil [5-FU] capecitabine, or S-1),
   * platinum (cisplatin or oxaliplatin),
   * taxanes (paclitaxel or docetaxel) or epirubicin,
   * irinotecan,
   * trastuzumab in case of human epidermal growth factor receptor 2 (HER2)-positive,
   * ramucirumab
   * nivolumab
   * pembrolizumab
5. Disease progression within 6 months after the last treatment.
6. Adequate bone-marrow, renal and liver function.
7. Eastern Cooperative Oncology Group (ECOG) performance status of ≤1.
8. Expected survival of ≥12 weeks, in the opinion of the investigator.

Exclusion Criteria:

1. History of another malignancy within 2 years prior to randomization except for the following: Bladder tumors considered superficial such as noninvasive (T1a) and carcinoma in situ (CIS); Curatively treated cervical CIS; Thyroid papillary cancer with prior treatment; Carcinoma of the skin without melanomatous features; Prostate cancer which had been surgically or medically treated and not likely to recur within 2 years.
2. Central nervous system (CNS) metastases as shown by radiology records or clinical evidence of symptomatic CNS involvement in the last 3 months prior to randomization.
3. Cytotoxic chemotherapy, surgery, immunotherapy, radiotherapy or other targeted therapies within 3 weeks (4 weeks in cases of ramucirumab, mitomycin C, nitrosourea, lomustine; 1 week in case of biopsy) prior to randomization (Adjuvant radiotherapy given to local area for non-curative symptom relief is allowed until 2 weeks before randomization.).
4. Therapy with clinically significant systemic anticoagulant or antithrombotic agents within 7 days prior to randomization that may prevent blood clotting and, in the investigator's opinion, could place the participant at risk.
5. Participants who had therapeutic paracentesis of ascites (>1 Liter [L]) within the 3 months prior to starting study treatment or who, in the opinion of the investigator, will likely need therapeutic paracentesis of ascites (>1L) within 3 months of starting study treatment.
6. Previous treatment with rivoceranib.
7. Known hypersensitivity to rivoceranib or components of the formulation.
8. Concomitant treatment with strong inhibitors or inducers of CYP3A4, CYP2C9, and CYP2C19.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 460 (Actual)
Dates: Start 2017-03-14 (Actual); Primary Completion 2019-02-15 (Actual); Study Completion 2020-09-23 (Actual)

CONTACTS AND LOCATIONS:
Locations (95):
- United States (5):
  - Mayo Clinic Phoenix, Scottsdale, Arizona
  - Highlands Oncology Group, Rogers, Arkansas
  - Karmanos Cancer Institute, Detroit, Michigan
  - Mayo Clinic Cancer Center, Rochester, Minnesota
  - Hudson Valley Cancer Centre, Hawthorne, New York
- France (5):
  - Centre Hospitalier Franco-Britannique; Oncologie Médicale, Levallois-Perret
  - Centre Leon-Berard (CLB), Lyon
  - Institut Regional du Cancer Montpellier (ICM), Montpellier
  - Centre Antoine-Lacassagne, Nice
  - Institut Gustave Roussy, Villejuif
- Germany (4):
  - Charite - Universitaetsmedizin Berlin - Medizinische Klinik mit Schwerpunkt Haematologie, Onkologie und Tumorimmunologie, Berlin
  - "Institut für Klinisch-Onkologische Forschung (IKF) Krankenhaus Nordwest gGmbH UCT - Universitäres Centrum für Tumorerkrankungen Frankfurt, Frankfurt
  - Facharztzentrum Eppendorf - Haematologisch-Onkologische Praxis Eppendorf (HOPE), Hamburg
  - Universitätsklinik Marburg, Klinik fur Innere Medizin, Schwerpunkt Haematologie, Onkologie und Immunologie, Marburg
- Italy (10):
  - Magna Graecia University- Department of Experimental and Clinical Medicine, Catanzaro
  - U.O Di Oncologia Ospedale Degli Infermi, Faenza
  - Fondazione IRCCS-Istituto Nazionale Tumori, Milan
  - Policlinico di Modena-Azienda Ospedaliero Universitaria di Modena.Oncologia ed Ematologia., Modena
  - Veneto Oncology Institute (IOV-IRCCS), Melanoma & Esophageal Oncology Unit, Padua
  - Ospedale di Piacenza - Oncology and heamatology, Piacenza
  - Ospedale "Felice Lotti", Pontedera
  - IRCCS/Arcispedale Santa Maria Nuova, Reggio Emilia
  - Rimini Hospital, Rimini
  - Ospedali Riuniti di Ancona - SOD Clinica Oncologica, Torrette
- Japan (15):
  - Hyogo Cancer Center, Hyōgo, Akasi-city
  - Chiba Cancer Center, Chiba, Chiba City
  - National Cancer Center Hospital, Tokyo, Chuo-ku
  - Kyushu University Hospital, Fukuoka, Higashi-ku
  - National Cancer Center Hospital East, Chiba, Kashiwa
  - St. Marianna University School of Medicine Hospital, Kanagawa, Kawasaki-shi
  - Saitama Cancer Center, Saitama, Kitaadachi-gun
  - Japan Community Health Care Organization Kyushu Hospital, Fukuoka, Kitakyushu-shi
  - The Cancer Institute Hospital of Japanese Foundation For Cancer Research, Tokyo, Koto-ku
  - National Hospital Organization Shikoku Cancer Center, Ehime, Matsuyama
  - Saku Central Hospital Advanced Care Center, Nagano, Saku-shi
  - Hokkaido University Hospital, Hokkaido, Sapporo
  - Keio University Hospital, Tokyo, Shinjuku-ku
  - Osaka University Hospital, Osaka, Suita
  - Aichi Cancer Center Hospital, Nagoya
- Poland (2):
  - Szpital Uniwersytecki w Krakowie, Odział Kliniczny Onkologii, Krakow
  - Centrum Onkologii-Instytut im. Marii Skłodowskiej-Curie, Klinika Gastroenterologii Onkologicznej, Warsaw
- Romania (4):
  - Saint Constantin Hospital (TEO HEALTH SA), Brasov
  - Institutul Oncologic "Prof. Dr. Ion Chiricuta" Cluj-Napoca, Sectia de Radioterapie I, Cluj-Napoca
  - S.C. Medisprof S.R.L., Cluj-Napoca
  - Centrul de Oncologie "Sf. Nectarie", Sectia de Oncologie Medicala, Craiova
- Russia (8):
  - State Budgetary Healthcare Institution of Arkhangelsk Region "Arkhangelsk Clinical Oncology Dispensary", Arkhangelsk
  - State Healthcare Institution "Kursk Regional Clinical Oncology Dispensary", Kursk
  - Omsk regional clinical oncology center, Omsk
  - Budgetary Healthcare Institution of Orel Region "Orel Oncology Dispensary", Oryol
  - State Budgetary Healthcare Institution of Stavropol Territory "Pyatigorsk Oncology Dispensary", Pyatigorsk
  - Federal State Budgetary Educational Institution of Higher Education "Academician I.P. Pavlov First St. Petersburg State Medical University" of the Ministry of Heaithcare of the Russian Federation, Saint Petersburg
  - Ogarev Mordovia State University, Saransk
  - State Budgetary Healthcare Institution "Republican Clinical Oncology Dispensary", Ufa
- South Korea (22):
  - Hallym University Sacred Heart Hospital, Anyang-si, Gyeonggi-do
  - National Cancer Center, Goyang-si, Gyeonggi-do
  - Ajou University Hospital, Suwon, Gyonggi-do
  - Inje University Haeundae Paik Hospital, Busan
  - Dong-A University Hospital, Busan
  - Pusan National University Hospital, Busan
  - Chungbuk National University Medical Center, Chuncheon
  - Kyungpook National University Medical Center, Daegu
  - Keimyung University Dongsan Medical Center, Daegu
  - Yeungnam University Medical Center, Daegu
  - Chungnam National University Hospital, Daejeon
  - Seoul National University Bundang Hospital, Gyeonggi-do
  - Gachon University Gil Medical Center, Incheon
  - Chungbuk National University Hospital, Jungbuk
  - Korea University Anam Hospital, Seoul
  - Severence Hospital, Yonsei University Health System, Seoul
  - Veterans Health Service (VHS) Medical Center, Seoul
  - ASAN Medical Center, Seoul
  - Gangnam Severance Hospital, Seoul
  - Samsung Medical Center, Seoul
  - Korea University Guro Hospital, Seoul
  - Ulsan University Hospital, Ulsan
- Taiwan (8):
  - Taipei Veterans General Hospital, Taipei, Beitou Dist
  - Chang Gung Memorial Hospital - Linko Branch, Taoyuan District, Kuei Shan Hsiang
  - Chi Mei Medical Center - LiouYing Branch, Tainan, Liuying DIst
  - Chang Gung Memorial Hospital - Kaohsiung Branch, Kaohsiung City, Niaosong Dist
  - Kaohsiung Medical University Hospital, Kaohsiung City, Sanmin Dist
  - China Medical University Hospital, Taichung, Taichung City
  - National CHeng Kung University Hospital, Tainan, Tainan City
  - National Taiwan University Hospital, Taipei, Zhongzheng Dist
- Ukraine (9):
  - Dnipropetrovsk Medical Academy, Department of Oncology, Dnipro
  - Communal Institution "Ivano-Frankivsk Regional Oncological Center", Ivano-Frankivsk
  - Communal Institution "Kharkiv Regional Clinical Oncology Center ", Chemotherapy department #1, Medical Academy of Postgraduate Education, Oncology and Pediatric Oncology, Kharkiv
  - Kherson Regional Oncological Dispensary, Kherson
  - Municipal Institution Kryvyi Rig Oncology Dispensary", Chemotherapy Department, Kryvyi Rih
  - Municipal Institution "Kyiv City Clinical Oncological Center", Kyiv
  - Communal Institution "Transcarpathian Regional Clinical Oncological Center", Uzhhorod
  - Communal Institution "Vinnytsia Regional Clinical Oncology Dispensary", Vinnytsia
  - State institution "Zaporizhzhia Medical Academy of Postgraduate Education MOH Ukraine", Department of oncology based on Municipal Institution "Zaporizhzhia Regional Clinical Oncology Dispensary" Zaporizhzhia Regional Assembly, Zaporizhzhia
- United Kingdom (3):
  - Royal Marsden Hospital London, London
  - The Christie NHS Foundation Trust, Manchester
  - Royal Marsden Hospital Surrey, Sutton

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants were randomized to receive either rivoceranib +best supportive care (BSC) or placebo +BSC for approximately 24 months. Participants who benefited from rivoceranib were permitted to continue rivoceranib during an extension period of the study, up to approximately 36 months. Participants in the extension period were followed for survival status only. Only participants whose reason for study discontinuation was death are included. See the AE module for All-Cause Mortality Deaths.
Groups:
- Rivoceranib Plus Best Supportive Care (BSC): Participants received rivoceranib 700 milligrams (mg) orally once per day during each cycle plus BSC. BSC is defined as palliative, non-cancer therapy. Each cycle duration was 28 days.
- Placebo Plus BSC; Extension Phase: Placebo Plus BSC: Participants received matching placebo to rivoceranib orally once per day during each cycle plus BSC. BSC is defined as palliative, non-cancer therapy. Each cycle duration was 28 days.
- Extension Phase: Rivoceranib Plus BSC: Participants received rivoceranib 700 mg orally once per day during each cycle plus BSC. BSC is defined as palliative, non-cancer therapy. Each cycle duration was 28 days.
Period: Core Phase
Arm/Group | Rivoceranib Plus Best Supportive Care (BSC) | Placebo Plus BSC | Extension Phase: Rivoceranib Plus BSC | Extension Phase: Placebo Plus BSC
Started | 308 | 152 | 0 | 0
Received at Least 1 Dose of Study Drug | 307 | 151 | 0 | 0
Completed | 52 | 28 | 0 | 0
Not Completed | 256 | 124 | 0 | 0
Not completed — Withdrawal by Subject | 13 | 4 | 0 | 0
Not completed — Death | 232 | 110 | 0 | 0
Not completed — Lost to Follow-up | 4 | 7 | 0 | 0
Not completed — Physician Decision | 7 | 2 | 0 | 0
Not completed — Study Closed | 0 | 1 | 0 | 0
Period: Extension Phase
Arm/Group | Rivoceranib Plus Best Supportive Care (BSC) | Placebo Plus BSC | Extension Phase: Rivoceranib Plus BSC | Extension Phase: Placebo Plus BSC
Started | 0 | 0 | 52 | 28
Completed | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 52 | 28
Not completed — Death | 0 | 0 | 34 | 16
Not completed — Lost to Follow-up | 0 | 0 | 1 | 1
Not completed — Study Closed | 0 | 0 | 17 | 11

BASELINE CHARACTERISTICS:
Population: The Intent to Treat (ITT) set consists of data from all participants who were randomized. In the ITT set, participants were included in the group to which they were randomized.
Groups:
- Total: Total of all reporting groups
Arm/Group | Rivoceranib Plus Best Supportive Care (BSC) | Placebo Plus BSC | Total
Number analyzed (Participants) | 308 | 152 | 460
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.03 (11.11) | 59.96 (10.63) | 60.01 (10.94)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 67 | 40 | 107
  Male | 241 | 112 | 353
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 0 | 5
  Not Hispanic or Latino | 303 | 152 | 455
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 207 | 105 | 312
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 100 | 46 | 146
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival (OS)
Description: OS was defined as the time from randomization to death. Participants alive or lost to follow-up at the end of study (EOS) were censored.
Time Frame: Day 1 (randomization) up to approximately 36 months
Population: The ITT set for the OS final analysis consisted of data from all participants who were randomized, including participants who were still in OS follow-up at the time of primary analysis. In the ITT set, participants were included in the group to which they were randomized.
Measure: Median (95% Confidence Interval); unit: Months
Groups:
- Rivoceranib Plus Best Supportive Care (BSC): Participants received rivoceranib 700 mg orally once per day during each cycle plus BSC. BSC is defined as palliative, non-cancer therapy. Each cycle duration was 28 days.
Arm/Group | Rivoceranib Plus Best Supportive Care (BSC) | Placebo Plus BSC
Number analyzed (Participants) | 308 | 152
Months | 5.82 [5.26 to 6.47] | 5.13 [4.47 to 6.24]

2. Secondary Outcome: Progression-free Survival (PFS) Per Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST 1.1)
Description: PFS was defined as the time from randomization to either documented radiological progression or death from any cause. Participants alive and free of progression at the EOS were censored.
Time Frame: Up to approximately 24 months
Population: The ITT set consisted of data from all participants who were randomized. In the ITT set, participants were included in the group to which they were randomized.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Rivoceranib Plus Best Supportive Care (BSC) | Placebo Plus BSC
Number analyzed (Participants) | 308 | 152
Months | 2.83 [2.07 to 3.52] | 1.77 [1.71 to 1.84]

3. Secondary Outcome: Objective Response Rate (ORR) Per RECIST 1.1
Description: ORR was defined as the percentage of participants in the analysis population with the best overall response of Complete Response (CR: disappearance of all target lesions and reduction in short axis of any nodal target lesions to <10 millimeter [mm]) or a Partial Response (PR: ≥30% decrease in the sum of the longest diameters of the target lesions, taking as a reference the baseline sum diameters) per RECIST 1.1.
Time Frame: Up to approximately 24 months
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Rivoceranib Plus Best Supportive Care (BSC) | Placebo Plus BSC
Number analyzed (Participants) | 308 | 152
Percentage of Participants | 6.5 [3.74 to 9.25] | 1.3 [0.16 to 4.67]

4. Secondary Outcome: Disease Control Rate (DCR)
Description: DCR was defined as the proportion of participants with a Best Overall Response of CR, PR, or stable disease (SD: Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as a reference the smallest sum diameter while on study) per RECIST 1.1.
Time Frame: Up to approximately 24 months
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Rivoceranib Plus Best Supportive Care (BSC) | Placebo Plus BSC
Number analyzed (Participants) | 308 | 152
Percentage of Participants | 40.3 [34.78 to 45.74] | 13.2 [7.78 to 18.53]

5. Secondary Outcome: Change From Baseline in Global Health Status/Quality of Life (QoL) Measured by European Organization for Research and Treatment of Cancer Quality of Life Questionnaire Core 30 (EORTC QLQ-C30)
Description: EORTC QLQ-C30 is a cancer specific Questionnaire with 30 questions for assessing the health-related QOL of cancer participants. The questionnaire incorporates 5 functional scales, 4 symptom scales, a global QOL scale, and single items for the assessment of additional systems commonly reported by cancer participants. All items are scored on 4-point Likert scales, ranging from 1 ('not at all') to 4 ('very much'), with the exception of 2 items in the global QOL scale which use modified 7-point linear analog scales. A linear transformation was used to standardize all scores and single-items to a scale of 0 to 100. For the functioning scales, a higher score indicated greater functioning and for the symptom scales, a higher score indicated a greater symptom burden.
Time Frame: Baseline, End of Treatment (EOT) (Up to 24 months)
Population: The ITT set consisted of data from all participants who were randomized. In the ITT set, participants were included in the group to which they were randomized. Overall number of participants indicates total number of participants with evaluable data.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Rivoceranib Plus Best Supportive Care (BSC) | Placebo Plus BSC
Number analyzed (Participants) | 207 | 99
units on a scale | -17.51 (22.72) | -18.01 (26.80)

6. Secondary Outcome: Change From Baseline in European Organization for the Research and Treatment of Cancer Quality of Life Questionnaire-Stomach Cancer Specific (EORTC QLQ-STO22) Score
Description: EORTC QLQ-STO22 is a 22-item gastric cancer-specific questionnaire-integrating system for assessing the health-related QOL of gastric cancer participants. Most questions use 4-point scale (1 'Not at all' to 4 'Very much'; 1 question was a yes or no answer). A linear transformation was used to standardize all scores and single-items to a scale of 0 to 100. For the functioning scales, a higher score indicates greater functioning and for the symptom scales, a higher score indicates a greater symptom burden.
Time Frame: Baseline, EOT (Up to 24 months)
Population: The ITT set consisted of data from all participants who were randomized. In the ITT set, participants were included in the group to which they were randomized. Overall number of participants indicates total at baseline, number of participants analyzed indicates number of participants with evaluable data.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Rivoceranib Plus Best Supportive Care (BSC) | Placebo Plus BSC
Number analyzed (Participants) | 207 | 99
units on a scale
  Body Image: number analyzed (Participants) | 205 | 99
  Body Image | 11.71 (29.95) | 9.43 (35.01)
  Dyspnea | 16.64 (26.34) | 16.50 (24.91)
  Pain | 12.72 (23.96) | 13.75 (21.91)
  Reflux Symptoms | 11.46 (24.80) | 8.31 (21.73)
  Eating Restrictions | 18.12 (26.45) | 17.76 (22.89)
  Anxiety | 13.69 (23.64) | 10.55 (26.91)
  Dry Mouth: number analyzed (Participants) | 207 | 98
  Dry Mouth | 20.77 (33.22) | 11.56 (29.15)
  Taste | 15.30 (32.46) | 14.48 (30.18)
  Hair Loss: number analyzed (Participants) | 206 | 99
  Hair Loss | -15.37 (33.71) | -18.69 (30.05)

7. Secondary Outcome: Change From Baseline in EuroQol 5-Dimension 5-Level Visual Analogue Scale (EQ-5D-5L VAS) Score
Description: EQ-5D-5L Questionnaire consists of EQ-5D-5L descriptive system and the visual analogue scale (VAS). The descriptive system comprises the 5 dimensions (mobility, self-care, usual activities, pain/discomfort, and anxiety/depression) and each dimension has 5 levels. The VAS is designed to rate the participant's current health state on a scale from 0 to 100, where 0 represents the worst imaginable health state and 100 represents the best imaginable health state.
Time Frame: Baseline, EOT (Up to 24 months)
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Rivoceranib Plus Best Supportive Care (BSC) | Placebo Plus BSC
Number analyzed (Participants) | 207 | 98
units on a scale | -18.48 (19.11) | -15.36 (21.61)

8. Secondary Outcome: Number of Participants Per QOL Dimension Response as Measured by the EuroQol 5-Dimension 5-Level (EQ-5D-5L) Questionnaire
Description: EQ-5D-5L Questionnaire comprises the 5 dimensions (mobility, self-care, usual activities, pain/discomfort, and anxiety/depression) and each dimension has 5 levels of response.
Time Frame: EOT (Month 24)
Population: The ITT set consisted of data from all participants who were randomized. In the ITT set, participants were included in the group to which they were randomized. Overall number of participants indicates total at baseline.
Measure: Count of Participants; unit: Participants
Arm/Group | Rivoceranib Plus Best Supportive Care (BSC) | Placebo Plus BSC
Number analyzed (Participants) | 308 | 152
Participants
  Mobility: No problems | 46 | 27
  Mobility: Slight problems | 60 | 27
  Mobility: Moderate problems | 51 | 23
  Mobility: Severe problems | 43 | 17
  Mobility: Unable | 8 | 6
  Mobility: Missing | 100 | 52
  Self Care: No problems | 100 | 54
  Self Care: Slight problems | 47 | 22
  Self Care: Moderate problems | 40 | 10
  Self Care: Severe problems | 14 | 7
  Self Care: Unable | 7 | 7
  Self Care: Missing | 100 | 52
  Usual Activities: No problems | 36 | 24
  Usual Activities: Slight problems | 61 | 36
  Usual Activities: Moderate problems | 56 | 18
  Usual Activities: Severe problems | 43 | 13
  Usual Activities: Unable | 12 | 9
  Usual Activities: Missing | 100 | 52
  Pain/Discomfort: No pain or discomfort | 25 | 13
  Pain/Discomfort: Slight pain or discomfort | 61 | 36
  Pain/Discomfort: Moderate pain or discomfort | 67 | 26
  Pain/Discomfort: Severe pain or discomfort | 47 | 19
  Pain/Discomfort: Extreme pain or discomfort | 8 | 6
  Pain/Discomfort: Missing | 100 | 52
  Anxiety/Depression: Not anxious or depressed | 49 | 26
  Anxiety/Depression: Slightly anxious or depressed | 60 | 36
  Anxiety/Depression: Moderately anxious or depressed | 62 | 25
  Anxiety/Depression: Severely anxious or depressed | 29 | 8
  Anxiety/Depression: Extremely anxious or depressed | 8 | 5
  Anxiety/Depression: Missing | 100 | 52

ADVERSE EVENTS:
Time Frame: Up to approximately 36 months
Description: The Safety set consisted of data from all participants in the ITT set who received at least 1 dose of rivoceranib or placebo. In the Safety set, participants were included in the group based on the treatment that was received. Safety data was analyzed by the Safety set which includes participants who were alive and on treatment or in OS follow-up. All-Cause Mortality includes deaths that led to study discontinuation and deaths that occurred during safety follow up.
Arm/Group | Rivoceranib Plus Best Supportive Care (BSC) | Placebo Plus BSC
All-Cause Mortality (participants affected / at risk) | 283/307 | 134/151
Serious Adverse Events (participants affected / at risk) | 149/307 | 66/151
Other Adverse Events (participants affected / at risk) | 299/307 | 140/151
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Rivoceranib Plus Best Supportive Care (BSC) (N=307) | Placebo Plus BSC (N=151)
Abdominal pain (Gastrointestinal disorders) | 15 | 3
Ileus (Gastrointestinal disorders) | 5 | 4
Vomiting (Gastrointestinal disorders) | 5 | 2
Gastric haemorrhage (Gastrointestinal disorders) | 4 | 2
Dysphagia (Gastrointestinal disorders) | 3 | 3
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 2 | 2
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 4 | 0
Obstruction gastric (Gastrointestinal disorders) | 3 | 2
Small intestinal obstruction (Gastrointestinal disorders) | 2 | 2
Asthenia (General disorders) | 8 | 8
Pyrexia (General disorders) | 6 | 1
Pain (General disorders) | 1 | 2
General physical health deterioration (General disorders) | 2 | 2
Cholangitis (Hepatobiliary disorders) | 2 | 4
Bile duct obstruction (Hepatobiliary disorders) | 5 | 0
Pneumonia (Infections and infestations) | 8 | 0
Decreased appetite (Metabolism and nutrition disorders) | 8 | 4
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 4 | 2
Ascites (Gastrointestinal disorders) | 3 | 1
Diarrhoea (Gastrointestinal disorders) | 3 | 0
Abdominal pain upper (Gastrointestinal disorders) | 2 | 1
Pancreatitis (Gastrointestinal disorders) | 3 | 0
Subileus (Gastrointestinal disorders) | 1 | 1
Gastric perforation (Gastrointestinal disorders) | 2 | 0
Gastric stenosis (Gastrointestinal disorders) | 1 | 1
Haematochezia (Gastrointestinal disorders) | 1 | 1
Large intestine perforation (Gastrointestinal disorders) | 2 | 0
Mechanical ileus (Gastrointestinal disorders) | 1 | 1
Stomatitis (Gastrointestinal disorders) | 2 | 0
Acute abdomen (Gastrointestinal disorders) | 1 | 0
Intestinal infarction (Gastrointestinal disorders) | 1 | 0
Abdominal distension (Gastrointestinal disorders) | 1 | 0
Enterocolitis (Gastrointestinal disorders) | 0 | 1
Haematemesis (Gastrointestinal disorders) | 0 | 1
Ileus paralytic (Gastrointestinal disorders) | 0 | 1
Intestinal obstruction (Gastrointestinal disorders) | 1 | 0
Large intestinal obstruction (Gastrointestinal disorders) | 1 | 0
Malignant dysphagia (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 1 | 0
Oesophageal pain (Gastrointestinal disorders) | 0 | 1
Oesophageal perforation (Gastrointestinal disorders) | 1 | 0
Oesophageal stenosis (Gastrointestinal disorders) | 1 | 0
Pancreatitis acute (Gastrointestinal disorders) | 1 | 0
Volvulus (Gastrointestinal disorders) | 1 | 0
Disease progression (General disorders) | 1 | 1
Fatigue (General disorders) | 1 | 0
Death (General disorders) | 0 | 1
Localised oedema (General disorders) | 1 | 0
Oedema peripheral (General disorders) | 0 | 1
Sudden death (General disorders) | 0 | 1
Hepatic failure (Hepatobiliary disorders) | 3 | 0
Jaundice cholestatic (Hepatobiliary disorders) | 2 | 1
Hyperbilirubinaemia (Hepatobiliary disorders) | 2 | 1
Biliary dilatation (Hepatobiliary disorders) | 2 | 0
Hepatic function abnormal (Hepatobiliary disorders) | 2 | 0
Cholecystitis (Hepatobiliary disorders) | 2 | 0
Hepatitis (Hepatobiliary disorders) | 0 | 1
Jaundice (Hepatobiliary disorders) | 1 | 0
Bile duct stenosis (Hepatobiliary disorders) | 1 | 0
Cholangitis acute (Hepatobiliary disorders) | 0 | 1
Cholecystitis acute (Hepatobiliary disorders) | 1 | 0
Liver disorder (Hepatobiliary disorders) | 0 | 1
Peritonitis (Infections and infestations) | 1 | 1
Septic shock (Infections and infestations) | 1 | 1
Biliary sepsis (Infections and infestations) | 2 | 0
Biliary tract infection (Infections and infestations) | 0 | 1
Endophthalmitis (Infections and infestations) | 1 | 0
Escherichia sepsis (Infections and infestations) | 1 | 0
Gastroenteritis (Infections and infestations) | 1 | 0
Oesophageal candidiasis (Infections and infestations) | 1 | 0
Urethritis (Infections and infestations) | 0 | 1
Hypernatraemia (Metabolism and nutrition disorders) | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0
Cachexia (Metabolism and nutrition disorders) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 0
Hyperuricaemia (Metabolism and nutrition disorders) | 1 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 0
Hypophagia (Metabolism and nutrition disorders) | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Posterior reversible encephalopathy syndrome (Nervous system disorders) | 2 | 0
Spinal cord compression (Nervous system disorders) | 1 | 1
Cerebral haemorrhage (Nervous system disorders) | 1 | 0
Cerebral infarction (Nervous system disorders) | 1 | 0
Epilepsy (Nervous system disorders) | 1 | 0
Haemorrhage intracranial (Nervous system disorders) | 0 | 1
Headache (Nervous system disorders) | 1 | 0
Paraesthesia (Nervous system disorders) | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 3 | 1
Nephropathy toxic (Renal and urinary disorders) | 0 | 1
Renal impairment (Renal and urinary disorders) | 1 | 0
Urinary retention (Renal and urinary disorders) | 0 | 1
Hydronephrosis (Renal and urinary disorders) | 0 | 1
Anaemia (Blood and lymphatic system disorders) | 3 | 2
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 1 | 1
Blood bilirubin increased (Investigations) | 2 | 0
Lipase increased (Investigations) | 2 | 0
Amylase increased (Investigations) | 1 | 0
Blood creatinine increased (Investigations) | 0 | 1
Gamma-glutamyltransferase increased (Investigations) | 0 | 1
Neutrophil count decreased (Investigations) | 1 | 0
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 3
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Acute myocardial infarction (Cardiac disorders) | 1 | 0
Cardiac failure (Cardiac disorders) | 1 | 0
Cardiac ventricular thrombosis (Cardiac disorders) | 1 | 0
Pericardial effusion (Cardiac disorders) | 0 | 1
Supraventricular tachycardia (Cardiac disorders) | 1 | 0
Ventricular fibrillation (Cardiac disorders) | 1 | 0
Subdural haemorrhage (Injury, poisoning and procedural complications) | 1 | 0
Intestinal anastomosis complication (Injury, poisoning and procedural complications) | 1 | 0
Radiation mucositis (Injury, poisoning and procedural complications) | 1 | 0
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 | 0
Subdural haematoma (Injury, poisoning and procedural complications) | 0 | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Spinal pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Delirium (Psychiatric disorders) | 1 | 0
Delusion (Psychiatric disorders) | 0 | 1
Adrenal insufficiency (Endocrine disorders) | 1 | 0
Device malfunction (Product Issues) | 0 | 1
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 | 0
Central venous catheter removal (Surgical and medical procedures) | 1 | 0
Deep vein thrombosis (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Rivoceranib Plus Best Supportive Care (BSC) (N=307) | Placebo Plus BSC (N=151)
Abdominal pain (Gastrointestinal disorders) | 78 | 30
Diarrhoea (Gastrointestinal disorders) | 92 | 22
Nausea (Gastrointestinal disorders) | 72 | 34
Stomatitis (Gastrointestinal disorders) | 69 | 5
Vomiting (Gastrointestinal disorders) | 53 | 21
Constipation (Gastrointestinal disorders) | 51 | 23
Abdominal pain upper (Gastrointestinal disorders) | 29 | 8
Dyspepsia (Gastrointestinal disorders) | 24 | 10
Ascites (Gastrointestinal disorders) | 15 | 13
Asthenia (General disorders) | 83 | 30
Fatigue (General disorders) | 77 | 16
Pyrexia (General disorders) | 36 | 17
Oedema peripheral (General disorders) | 18 | 5
Decreased appetite (Metabolism and nutrition disorders) | 132 | 45
Hypoalbuminaemia (Metabolism and nutrition disorders) | 34 | 16
Aspartate aminotransferase increased (Investigations) | 71 | 11
Weight decreased (Investigations) | 69 | 12
Alanine aminotransferase increased (Investigations) | 64 | 9
Blood alkaline phosphatase increased (Investigations) | 43 | 13
Platelet count decreased (Investigations) | 46 | 6
Blood bilirubin increased (Investigations) | 37 | 8
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 81 | 6
Rash (Skin and subcutaneous tissue disorders) | 19 | 4
Hypertension (Vascular disorders) | 106 | 5
Anaemia (Blood and lymphatic system disorders) | 64 | 41
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 44 | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 16 | 12
Headache (Nervous system disorders) | 41 | 5
Back pain (Musculoskeletal and connective tissue disorders) | 17 | 8
Insomnia (Psychiatric disorders) | 18 | 10
Proteinuria (Renal and urinary disorders) | 90 | 11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2018-11-16): https://cdn.clinicaltrials.gov/large-docs/11/NCT03042611/Prot_000.pdf
  • Statistical Analysis Plan (2019-02-01): https://cdn.clinicaltrials.gov/large-docs/11/NCT03042611/SAP_001.pdf